CLINICAL TRIAL: NCT01528033
Title: Treatment of Subcutaneous Abdominal Wound Healing Impairment After Surgery Without Fascial Dehiscence by Vacuum Assisted Closure™(SAWHI-V.A.C.® Study) Versus Standard Conventional Wound Therapy
Brief Title: Treatment Study of Vacuum Assisted Closure for Postsurgical Subcutaneous Abdominal Wound Healing Impairments
Acronym: SAWHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: KCI Europe Holding B.V. (Industry)
Responsible Party: Principal Investigator, Doerthe Seidel, Interim Scientific Leader of the Centre for Clinical Trials and Innovation, University of Witten/Herdecke
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VAC2010-56; 00000648 (Registry Identifier: DRKS)
Record Dates: First submitted 2012-02-02; First posted 2012-02-07 (Estimated); Results first posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Wound Healing Disorder; Impaired Wound Healing; Abdominal Wound Healing Disorder; Abdominal Wound Healing Impairment; Acute Postsurgical Subcutaneous Wound
Keywords: surgical wound; wound healing disorder; Wound healing impairment; post surgical wound healing disorder; abdominal wound healing impairment; Vacuum Assisted Closure; negative pressure wound therapy
MeSH Terms: conditions — Surgical Wound | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vacuum Assisted Closure® (Experimental): Negative pressure wound therapy
  Interventions: Device: Vacuum Assisted Closure®
- Standard conventional wound therapy (Active Comparator): According to institutional clinical standards
  Interventions: Other: Standard conventional wound therapy

INTERVENTIONS:
Device: Vacuum Assisted Closure® — Vacuum Assisted Closure® (V.A.C.®) Therapy within a maximum study treatment time of 42 days.
  VAC® Therapy Systems used within the trial are ActiV.A.C.®, InfoV.A.C.®, V.A.C. Freedom®, V.A.C. Via® and VAC Ulta®. All used systems are equally eligible for the treatment of subcutaneous abdominal wounds and should be used according to availability and local preferences within the trial site.
  Systems differ regarding user surface and display and processing of data. For the treatment of subcutaneous abdominal wounds the V.A.C.® Granufoam Dressing (size medium and big) is recommended.
  Other Names: Negative Pressure Wound Therapy
  Arms: Vacuum Assisted Closure®
Other: Standard conventional wound therapy — Standard conventional wound therapy (SCWT) according to institutional clinical standards within a maximum study treatment time of 42 days
  Arms: Standard conventional wound therapy

SUMMARY:
This clinical study is performed in several German, Dutch and Belgian hospitals to evaluate the efficacy of Vacuum Assisted Closure® (V.A.C.®) for the treatment of postsurgical abdominal wound healing impairments after surgery. Therefore the underlying layer of fibrous tissue that permeates the internal organs must be intact.

Main outcome measure is the time until complete wound closure that sustained for a minimum of 14 days. Furthermore the therapy options will be examined regarding several other clinical, safety, patient reported and economic parameters.

Patients will be assigned equally and by chance to both treatment groups. Study participants as well as the attending doctors and nurses will be informed about the assignment to the respective treatment arm.

The primary outcome measure and some of the secondary parameters like reappearance of the wound and the development of the wound size over time, examined within an active study treatment time of 42 days, will be photographed and analysed under the use of a central computer system. The central analysing personal will not be informed about patient details or therapy allocation.

Patients with at first closed belly wounds with wound healing disorder in the postoperative course after surgery without an opening of the underlying layer of fibrous tissue are eligible to be included in the trial if the diagnosis of a wound healing impairment in the postoperative course is manifested as a wound with spontaneous dehiscence, a wound that requires an active reopening of the suture by the treating physician or a wound that cannot be closed by primary intention and requires further treatment to achieve permanent closure.

Study participants will be selected and enrolled within clinical surgical departments which provide the respective personal, structural and scientific background for the conduction of the trial project.

Trial therapy will be started in-hospital and may be continued in ambulatory care. It is very important to examine the therapy options also in the ambulant care setting thus study participants with good health who are able to continue the specific wound treatment in ambulant should be transferred to the ambulant service as soon as possible.

DETAILED DESCRIPTION:
The Institute for Research in Operative Medicine as part of the Private University of Witten /Herdecke is planning and performing a clinical trial project to evaluate the efficacy of Vacuum Assisted Closure® (V.A.C.®) Therapy for the treatment of postsurgical abdominal wound healing impairments after surgery without fascial dehiscence. The clinical trial project is fully financed by Kinetic Concepts Incorporated (KCI). The V.A.C.® Therapy devices that will be used in this study include the ActiV.A.C.® Therapy System, InfoV.A.C.® Therapy System, and V.A.C. Freedom® Therapy System. All V.A.C.® Therapy devices to be utilized in this study bear the CE mark and will be operated within normal conditions of use and according to manufacturer's specifications.

Background of the clinical trial project is the decision of the Joint Federal Committee of Germany (Gemeinsamer Bundesausschusses (G-BA)) that Vacuum assisted closure therapy is inadmissible to be a standard benefit of health insurance companies in Germany.

This decision is based on systematic review & meta-analysis of existing trials performed by Institute for Quality and Economic Efficiency in the Healthcare System (Institut für Qualität und Wirtschaftlichkeit im Gesundheitswesen (IQWiG)) which showed an insufficient state of evidence regarding the efficacy of negative pressure wound therapy for the treatment of acute and chronic wounds.

This study project compares Vacuum Assisted Closure® and standard conventional wound therapy in the treatment of acute abdominal wounds after surgery without fascial dehiscence and will be conducted in abdominal surgical hospital departments with the required structural, manpower, and scientific qualifications. Patients will be stratified according to hospital and wound size. Trial therapy will be started in-hospital and may be continued in ambulatory care.

The study is designed as a multinational, multicentre, prospective randomized controlled, adaptive design, clinical superiority trial, with blinded photographic analysis of the primary endpoint.

The primary objective is to compare the clinical, safety, and economic outcomes of V.A.C.® Therapy and SCWT in postsurgical abdominal wound healing impairments without fascial dehiscence.

The primary outcome to be observed in this study is time to complete abdominal wound closure where closure is observed at or before day 42 and is confirmed to have been sustained for a period of at least 14 consecutive days. This study design also will allow detailed description of specific covariates to determine their effect on response variables (healing).

This study's hypothesis is that the use of the V.A.C.® Therapy System, when compared to SCWT in the management of post-surgical abdominal wound healing impairments with intact fascia, will result in a decrease in the time to achieve complete wound closure with confirmation after subsequent 14 days.

Using V.A.C.® Therapy is an effective and safe treatment option for hospitals as well as for outpatient care for treatment of subcutaneous abdominal wounds with wound healing impairment in the postoperative course.

Randomisation to treatment arms will be performed at a 1:1 ratio. Randomisation will be performed via a centralized system with an Internet-based tool. To address issues of blinding, wound photo documentation will be obtained during the trial and confirmation of wound closure will be assessed via blinded photographic analysis, which will serve as the method of primary endpoint analysis.

Primary closed abdominal wounds with wound healing disorder in the postoperative course after surgical intervention without fascial dehiscence are eligible to be included in the trial if the diagnosis of a wound healing impairment in the postoperative course is manifested as a wound with spontaneous dehiscence, a wound that requires an active reopening of the suture by the treating physician or a wound that cannot be closed by primary intention and requires further treatment to achieve permanent closure.

During active recruitment phase, the pre-trial estimates indicate approximately 600 patients will be required to yield the target of 552 evaluable participants. Using an adaptive design study sample-size calculations will be re-estimated upon planed interim analysis of study data of 250 patients. Patients will be enrolled from approximately 25 centres in Germany, the United Kingdom, Belgium and the Netherlands.

The evaluation of the primary Endpoint defined as time (number of days) to achieve complete wound closure verified by photo documentation and blinded, computer-based wound quality assessment as well as wound closure confirmation after 14 consecutive days and secondary endpoints including clinical endpoints like recurrences, safety endpoints, patient reported outcome parameters and economic-based outcome measures will provide data regarding efficacy and efficiency of NPWT therapy for the treatment of acute post-surgical abdominal wound healing impairment in hospital as well as in the ambulant setting.

The results of the study will be provided to make a contribution to the final decision of the Joint Federal Committee about NPWT to be a standard benefit of health insurance companies in Germany for inpatient and / or outpatient care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Post-surgical subcutaneous abdominal wound healing impairment
* Minimum wound size eligible for the application of the randomized treatment- Inclusion, randomization, adequate wound pre-treatment (Debridement) and start of therapy within 48 hours after reopening of the wound, diagnosis for nonclosable wound or in case of spontaneous wound dehiscence

Exclusion Criteria:

* Age < 18
* Noncompliance with study procedures, visit schedule and follow up
* Pregnancy
* Present or nonclosable defect of the abdominal fascia
* Any pre-existing or ongoing organ system failure, that cannot be stabilized or solved by appropriate medical treatment
* Necrotic tissue with eschar present
* Non-enteric and unexplored fistulas
* Malignancy of the wound
* Use of any other device based on the principle of negative pressure wound therapy on the study wound within ≤ 8 days prior to screening
* Competing therapies or procedures
* Simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doerthe Seidel, Principal Investigator — Witten / Herdecke University
Locations (15):
- Belgium (2):
  - UZ Brussel, Brussels
  - Department of Abdominal Surgery Gasthuisberg University Hospital, Leuven
- Germany (13):
  - Sana Klinikum Lichtenberg (Berlin), Berlin
  - Unfallkrankenhaus Berlin Klinik für Allgemein- und Viszeralchirurgie, Berlin
  - St. Josef-Hospital gGmbH Universitätsklinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum des Saarlandes, Klinik für Allgemeine Chirurgie, Viszeral-, Gefäß- und Kinderchirurgie, Homburg
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität, Mainz
  - Universitätsmedizin Mannheim Medizinische Fakultät Mannheim der Universität Heidelberg Chirurgische Klinik, Mannheim
  - Chirurgische Klinik und Poliklinik, Klinikum rechts der Isar, München
  - Ruppiner Kliniken GmbH, Neuruppin
  - Klinikum Ernst von Bergmann, Klinik für Allgemein- und Visceralchirurgie, Potsdam
  - Diakoniekrankenhaus Rotenburg, Rotenburg (Wümme)
  - Thüringen-Kliniken "Georgius Agricola" GmbH, Saalfeld
  - GRN-Klinik Sinsheim, Allgemein- und Viszeralchirurgie, Sinsheim

REFERENCES:
- [Background] Seidel D, Lefering R, Neugebauer EA. Treatment of subcutaneous abdominal wound healing impairment after surgery without fascial dehiscence by vacuum assisted closure (SAWHI-V.A.C.(R)-study) versus standard conventional wound therapy: study protocol for a randomized controlled trial. Trials. 2013 Nov 20;14:394. doi: 10.1186/1745-6215-14-394. PMID 24252551
- [Result] Seidel D, Diedrich S, Herrle F, Thielemann H, Marusch F, Schirren R, Talaulicar R, Gehrig T, Lehwald-Tywuschik N, Glanemann M, Bunse J, Huttemann M, Braumann C, Heizmann O, Miserez M, Kronert T, Gretschel S, Lefering R. Negative Pressure Wound Therapy vs Conventional Wound Treatment in Subcutaneous Abdominal Wound Healing Impairment: The SAWHI Randomized Clinical Trial. JAMA Surg. 2020 Jun 1;155(6):469-478. doi: 10.1001/jamasurg.2020.0414. PMID 32293657
- [Derived] Seidel D; SAWHI study group. Ambulatory negative pressure wound therapy of subcutaneous abdominal wounds after surgery: results of the SAWHI randomized clinical trial. BMC Surg. 2022 Dec 12;22(1):425. doi: 10.1186/s12893-022-01863-x. PMID 36503505
- See also: Sponsor — http://www.uni-wh.de

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled betweenAugust 2, 2011, and January 31, 2018 in 34 abdominal surgical departments of hospitals in Germany, Belgium, and the Netherlands
Groups:
- Vacuum Assisted Closure®: Negative pressure wound therapy
  Vacuum Assisted Closure®: Vacuum Assisted Closure® (V.A.C.®) Therapy within a maximum study treatment time of 42 days.
  VAC® Therapy Systems used within the trial are ActiV.A.C.®, InfoV.A.C.®, V.A.C. Freedom®, V.A.C. Via® and VAC Ulta®. All used systems are equally eligible for the treatment of subcutaneous abdominal wounds and should be used according to availability and local preferences within the study site.
  Systems differ regarding user surface and display and processing of data. For the treatment of subcutaneous abdominal wounds the V.A.C.® Granufoam Dressing (size medium and big) is recommended.
Period: Primary Endpoint Assessment ITT
Arm/Group | Vacuum Assisted Closure® | Standard Conventional Wound Therapy
Started | 273 | 266
Completed | 256 | 251
Not Completed | 17 | 15
Not completed — Withdrawal by Subject | 8 | 7
Not completed — No or deliquent informed consent | 3 | 3
Not completed — Death | 2 | 2
Not completed — Physician Decision | 2 | 1
Not completed — No post baseline documentation | 2 | 2
Period: Follow Up
Arm/Group | Vacuum Assisted Closure® | Standard Conventional Wound Therapy
Started | 256 | 251
Completed | 210 | 207
Not Completed | 46 | 44
Not completed — No data available | 46 | 44

BASELINE CHARACTERISTICS:
Population: Intention To Treat Population
Groups:
- NPWT: Negative Pressure Wound Therapy
- SCWT: Standard Conventional Wound Treatment
- Total: Total of all reporting groups
Arm/Group | NPWT | SCWT | Total
Number analyzed (Participants) | 256 | 251 | 507
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 64 (14) | 64 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 119 | 220
  Male | 155 | 132 | 287
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 245 | 241 | 486
  Netherlands | 2 | 1 | 3
  Belgium | 7 | 9 | 16
Weight [Mean (Standard Deviation); unit: Kilogram] | 86 (19) | 84 (21) | 85 (20)
Height [Mean (Standard Deviation); unit: Centimeters] | 172 (11) | 169 (11) | 171 (11)
BMI [Mean (Standard Deviation); unit: kg/m²] | 28.71 (8.58) | 29.5 (10.2) | 29.4 (8.4)
Smoking [Count of Participants; unit: Participants] | 65 | 55 | 120
Alcohol use [Count of Participants; unit: Participants] — Population: Only for those patientes with information available
  Participants
    number analyzed (Participants) | 255 | 250 | 505
    (all) | 111 | 114 | 225
Drug use [Count of Participants; unit: Participants] | 3 | 3 | 6
Nutritional status [Count of Participants; unit: Participants]
  Well nourished | 235 | 222 | 457
  Moderately or suspected of being malnourished | 18 | 26 | 44
  Severely malnourished | 3 | 3 | 6
Wound volume [Count of Participants; unit: Participants] — Population: Only for those patients with available Information
  Participants
    number analyzed (Participants) | 256 | 249 | 505
    <=60 cm*3 | 149 | 142 | 291
    >60 cm*3 | 107 | 107 | 214
Coagulation: Prothrombin Time (PT) [Mean (Standard Deviation); unit: percentage (%)] — Population: Laboratory values are only available for patients with blood samples collected within clinical routine
  percentage (%)
    number analyzed (Participants) | 149 | 148 | 297
    (all) | 88.3 (16.2) | 88.3 (17.8) | 88.3 (17.0)
Coagulation: International Normalized Ratio (INR) [Mean (Standard Deviation); unit: ratio] — Population: Laboratory values are only available for patients with blood samples collected within clinical routine
  ratio
    number analyzed (Participants) | 145 | 145 | 290
    (all) | 1.1 (0.2) | 1.1 (0.2) | 1.1 (0.2)
Coagulation: Partial Thromboplastin Time (pTT) [Mean (Standard Deviation); unit: seconds (s)] — Population: Laboratory values are only available for patients with blood samples collected within clinical routine
  seconds (s)
    number analyzed (Participants) | 146 | 146 | 292
    (all) | 33.9 (10.8) | 32.5 (10.4) | 33.2 (10.6)
Diagnosis of abdominal wound healing disorder [Count of Participants; unit: Participants]
  Spontaneous dehiscence | 57 | 52 | 109
  Active reopening | 198 | 193 | 391
  Wound left open after surgery | 2 | 9 | 11
Clinical signs of infection during screening [Count of Participants; unit: Participants] — Population: Only for those patients with Information available
  Participants
    No: number analyzed (Participants) | 256 | 250 | 506
    No | 122 | 116 | 238
    Not assesable: number analyzed (Participants) | 256 | 250 | 506
    Not assesable | 29 | 24 | 53
    Yes: number analyzed (Participants) | 256 | 250 | 506
    Yes | 105 | 110 | 215
Leven of surgical site infection according to CDC classification at Screening [Count of Participants; unit: Participants] — Population: Only for those patients with signs of clinical infection during Screening (NPWT=105; SCWT=110) and documentation availabe (NPWT=104; SCWT=110)
  Participants
    number analyzed (Participants) | 104 | 110 | 214
    Superficial incisional | 65 | 67 | 132
    Deep incisional | 37 | 39 | 76
    Organ or space infection | 2 | 4 | 6
Clinical signs of local infection at randomization, [Count of Participants; unit: Participants] — Population: Patients with documentation availabe at Randomization = 247
  Participants
    number analyzed (Participants) | 247 | 245 | 492
    No | 133 | 130 | 263
    Not assessable | 39 | 36 | 75
    Yes | 75 | 79 | 154
Level of surgical site infection according to CDC classification at Randomization [Count of Participants; unit: Participants] — Population: Only availabe for those patients with clinical signs of local infection during randomization (NPWT=75; SCWT=79) and documentation available (NPWT=73; SCWT=79)
  Participants
    number analyzed (Participants) | 73 | 79 | 152
    Superficial incisional | 43 | 43 | 86
    Deep incisional | 28 | 34 | 62
    Organ or space infection | 2 | 2 | 4
Main procedure that caused the abdominal wound healing impairment [Count of Participants; unit: Participants] — Population: Only for those patients with documentation available (NPWT=255; SCWT=248)
  Participants
    number analyzed (Participants) | 255 | 248 | 503
    Incision, excision, resection and anastomose of th | 94 | 93 | 187
    Other operations on the small and large intestine | 35 | 30 | 65
    Appendix surgery | 14 | 13 | 27
    Rectal surgery | 22 | 20 | 42
    Anal surgery | 0 | 0 | 0
    Esophagus surgery | 0 | 2 | 2
    Gastric incision, excision, and resection | 6 | 4 | 10
    Extended gastric resection and other gastric surge | 3 | 0 | 3
    Liver surgery | 8 | 8 | 16
    Gall bladder and bile ducts surgery | 23 | 17 | 40
    Pancreatic surgery | 13 | 11 | 24
    Closure of abdominal hernias | 18 | 13 | 31
    Operations on other abdominal regions | 15 | 27 | 42
    Other | 4 | 10 | 14

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Wound Closure
Description: Time (number of days) to achieve complete wound closure verified by photo documentation and blinded, computer-based wound quality assessment as well as wound closure confirmation after 14 consecutive days (14 days -0 / + 3)
  Complete wound closure is defined as:
  100% epithelialization No drainage from the wound No need for adjuvant therapy or dressing No presence of sutures
Time Frame: 42 days
Population: Intention To Treat Population
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | NPWT | SCWT
Number analyzed (Participants) | 256 | 251
Days | 36.1 [35.0 to 37.2] | 39.1 [38.3 to 40.0]

2. Secondary Outcome: Incidence of Confirmed and Verified Wound Closure
Description: Incidence of confirmed and verified wound closure achieved after a maximum study observation / treatment period of 42 days (+ 14 days to observe sustained closure)
Time Frame: 42 days
Population: Intention To Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | NPWT | SCWT
Number analyzed (Participants) | 256 | 251
Participants | 92 | 54

3. Secondary Outcome: Recurrence
Description: Recurrence of wound opening after confirmed wound closure
Time Frame: 132 days
Population: Intention To Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | NPWT | SCWT
Number analyzed (Participants) | 256 | 251
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 42 days for Adverse Events (AEs) and unsustained wound closures 132 days for Serious Adverse Events (SAEs)
Description: Mortality is presented for the ITT Population (NPWT N=256; SCWT N=251). AEs and SAEs were only collected if treatment-related. NPWT-, SCWT- and wound-related AEs were analyzed based on the Therapy Compliant (TC) population (study participants without unauthorized treatment changes) (N total NPWT=234; N total SCWT=201).This enables a clear assignment of the adverse event to one of the two treatment methods for study participants who actually received the randomized therapy.
Arm/Group | NPWT | SCWT
All-Cause Mortality (participants affected / at risk) | 24/256 | 15/251
Serious Adverse Events (participants affected / at risk) | 22/234 | 12/201
Other Adverse Events (participants affected / at risk) | 41/234 | 22/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPWT (N=234) | SCWT (N=201)
Adverse Device Events (NPWT-related) (Surgical and medical procedures) | 0 (0) | 0 (0)
Conventional Wound Treatment-related (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Wound-related (Skin and subcutaneous tissue disorders) | 22 (29) | 12 (12)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPWT (N=234) | SCWT (N=201)
Adverse Device Events (NPWT-related) (Surgical and medical procedures) | 13 (23) | 0 (0)
Conventional Wound Treatment - related (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Wound-related (Skin and subcutaneous tissue disorders) | 41 (51) | 22 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-17): https://cdn.clinicaltrials.gov/large-docs/33/NCT01528033/Prot_SAP_000.pdf